CLINICAL TRIAL: NCT00954837
Title: Utility of a Second Ultrasound-guided Fine Needle Aspiration for the Detection of Thyroid Cancer in the Management of Single Thyroid Nodules or Multinodular Goitre.
Brief Title: Assessment of Repeat Fine Needle Aspiration (FNA) to Detect Thyroid Cancer
Acronym: CYT2THYR
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: administrative delays too long
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ID RCB 2008-A00839-46
Record Dates: First submitted 2009-07-30; First posted 2009-08-07 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2013-05

CONDITIONS: Thyroid Cancer
Keywords: Thyroid cancer; thyroid FNA; repeat FNA; thyroid screening; thyroid ultrasonography; FNA screening
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Biopsy, Fine-Needle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fine needle aspiration (Other): Patient with solid nodules more than 10 mm in diameter will be biopsied by ultrasound-guided fine-needle aspiration(FNA)after consultation with an endocrinologist or ENT specialist.
  Interventions: Procedure: Fine needle aspiration

INTERVENTIONS:
Procedure: Fine needle aspiration — Classical needle biopsy techniques will be used, with patients lying on their backs with their necks in hyperextension. An initial ultrasound scan will be used to determine the site or sites at which the needle should be inserted. Following extensive disinfection of the skin of the neck, the needle will be inserted under ultrasound guidance. The needle will be moved gently backwards and forwards and displaced radially in a clockwise direction to recover cellular material by capillarity. In general, several (two or three) passages of the needle are required for a given nodule. It is possible to carry out FNA on up to three nodules in a single session. For each passage, a new, sterile, single-use needle will be used. The insertion of each needle will be preceded by an ultrasound scan.
  Other Names: Fine needle aspiration under ultrasonography

SUMMARY:
Thyroid nodules are common (prevalence of 12.7% in women), but are malignant in only 5% of cases. International experts agree that a preliminary cytological examination by fine needle aspiration (FNA) is required. The management of patients with cytological results consistent with malignant or suspicious for malignancy nodules is well codified and generally involves surgery. However, there is no consensus concerning 1) the utility of a second FNA during the monitoring of benign nodules. Certain studies have recommended a second FNA, whereas others have recommended ultrasound monitoring alone; 2) the contribution of ultrasound criteria to the decision as to whether to carry out a second FNA, particularly if the nodule increases in size; 3) the management of nodules classified as doubtful or suspect on needle biopsy, many of which prove to be benign (20 to 30% are malignant), raising questions about the utility of systematic thyroid surgery or the justification for a second FNA; 4) the management of patients with non significant (NS) findings on FNA, for whom immediate surgery, monitoring or a second FNA may be recommended and 5) the procedure to be followed for nodules present in patients with multinodular thyroid disease.

DETAILED DESCRIPTION:
Background :

A few studies have tried to evaluate the value of a second needle biopsy. Ultrasound criteria for malignancy have been described but are mostly unvalidated. Only a very small number of immunocytochemical studies using several antibodies have been reported, mostly dealing with series of less than 50 cases. The Bethesda State of Science Conference held in October 2007 (ahead on print, 2009) on fine-needle biopsy of the thyroid considered that no sufficiently robust studies of this technique had yet been carried out and that prospective studies were required.

Objectives:

The principal objective of this study is to determine the utility of a second needle biopsy in the routine management of patients presenting, for a given nodule, initial cytological results that were non-significant, benign, doubtful or suspect. The secondary objectives are to determine the utility of various pre-determined ultrasound criteria and of the collection of cells in liquid medium combined with immunocytochemistry.

Methodology:

Prospective study on a cohort of 400 patients attending consultations in the Internal Medicine/Endocrinology Department or the ENT Department, or referred by external doctors, whether working in hospitals or in private practice, participating in a protocol of single or multiple thyroid nodule disease assessment. Each patient will attend at least one consultation and undergo at least one thyroid ultrasound scan with fine-needle aspiration (FNA). Based on the result of this first needle biopsy, management will be oriented towards immediate surgery or follow-up for 6/12 or 18 months, with a second thyroid needle biopsy within a maximum of 18 months of follow-up.

Inclusion period: 18 months Duration of follow-up: up to18 months Total duration of the study: 36 months

Description of the techniques used in this protocol:

Radiological techniques :

They will then undergo ultrasound-guided fine-needle aspiration (FNA). Classical needle biopsy techniques will be used, with patients lying on their backs with their necks in hyperextension. An initial ultrasound scan will be used to determine the site or sites at which the needle should be inserted. Following extensive disinfection of the skin of the neck, the needle will be inserted under ultrasound guidance. The needle will be moved gently backwards and forwards and displaced radially in a clockwise direction to recover cellular material by capillarity. The material recovered will be diluted in 30 ml of CYTOLYT (Hologic), a transport medium for the recuperation of cells in liquid media. In general, several (two or three) passages of the needle are required for a given nodule. It is possible to carry out FNA on up to three nodules in a single session. For each passage, a new, sterile, single-use needle will be used. The insertion of each needle will be preceded by an ultrasound scan.

Surgical technique:

For all nodules for which surgery is indicated, LOBOISTHMECTOMY will be carried out with frozen sections (FS). There are three possibilities: 1) FS provides evidence of thyroid cancer. In such cases, total thyroidectomy is carried out, with dissection of the lymph nodes areas in the central (zone VI) and lateral (zones II to IV) zones on each side; 2) FS provides no evidence of malignancy. In such cases, the surgical intervention is limited to LOBOISTHMECTOMY; 3) FS shows the nodule in question to be suspect. In such cases, total thyroidectomy is not carried out before the definitive pathological results are known. It is widely accepted that recurrent dissection should also be carried out during this initial surgery. Indeed, if the definitive pathological examination shows the nodule to be cancerous, repeat surgical interventions with recurrent dissection are potentially much more damaging to the recurrent nerve.

If there is an indication for total thyroidectomy due to the presence of multiple nodules or multinodular goitre, FS is carried out for the entire thyroid, with sampling directed by the pathologist to determine whether central and lateral zone dissection should be carried out.

The sampling circuit :

All solid nodules more than 10 mm in diameter will be biopsied by FNA if there is only one such nodule or if there are no more than three such nodules. Only the largest nodule and nodules with suspect characteristics on ultrasound will be controlled by FNA if there are more than three nodules exceeding 10 mm in diameter. The procedure adopted depends on the individual nodule. Decisions concerning surgery are based on the most severe diagnosis obtained if several nodules are assessed.

For each nodule subjected to FNA, a complete radiological description will be written, regardless of the time-point at which the investigation is carried out (T0, T6, T12 or T18). For patients seen on several occasions during the study, any changes in one or several nodules observed on ultrasound scan will be noted.

The material collected by FNA will be deposited in liquid medium (Hologic; LBC technique). If several nodules are examined, the material from each nodule will be placed in a separate, clearly identified flask.

A complementary immunocytological study will be systematically carried out for all nodules other than those considered "benign and with no radiological modifications." If there is sufficient residual cell material, a panel of antibodies will be used, constituted from the available antibodies against the following: HBME1, cytokeratin 19, TTF1, thyrocalcitonin, thyroglobulin, CD3, CD20. The results will be delivered in two lots: first the cytological and morphological results alone, according to NCI Bethesda 2008 classification criteria, and then the immunocytochemical results, broken down into three categories (probably benign, probably malignant and inconclusive).

Potential implication :

The aim of the study is to intend clinical, radiological, cytological and surgical feasible recommendations for an accurate follow-up of benign single thyroid nodules or multinodular goiter. Thyroid nodules are essentially benign lesions ; therefore the main objective is to detect all the cancers but not to induce unnecessary surgical controls.

ELIGIBILITY:
Inclusion Criteria:

* Patient are more than 18 years old
* Patient with a unique or several thyroid solid nodules more than 10 mm wide
* Patient who accept to be followed over 18 months
* Study Informed patient, non opposed to his/her own data analyzes

Exclusion Criteria:

* Pregnant women
* Patient with previous data of thyroid cancer
* Patient with low TSH (inferior to local norm)
* Patient refusing thyroid surgery policy/ rule
* Irresponsible patient or patient refusing to participate
* Patient with clinical or psychological state not permitting study sample

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-04; Primary Completion 2011-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Status nodule | Inclusion, 6, 12 and 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Marie LALOI-MICHELIN, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris